CLINICAL TRIAL: NCT01862653
Title: Acupuncture for Sleep Disturbances in OEF/OIF Veterans With Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMCSD.2012.0053; HT9404-12-1-TS15(N12-P15) (Other Grant/Funding Number: Tri Service Nursing Research Program)
Record Dates: First submitted 2013-05-06; First posted 2013-05-24 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Post Traumatic Stress Disorder; Sleep Disturbance
Keywords: Post Traumatic Stress Disorder; Sleep Disturbance; Acupuncture
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Auricular Acupuncture (Experimental): An insomnia auricular acupuncture protocol will be administered for 30 minutes, three times per week, for three weeks in the intervention group.
  Interventions: Device: Auricular Acupuncture
- Control (No Intervention): The control group is a wait-list control group and will be offered the auricular acupuncture intervention after the study is complete. No intervention will be performed on control group.

INTERVENTIONS:
Device: Auricular Acupuncture — Subjects receiving the auricular acupuncture intervention will be treated in a quiet private room sitting in a comfortable chair. The external ear cartilage of both ears will be cleaned with isopropyl alcohol swabs. A clean insertion technique will be used with stainless steel SEIRIN D type acupuncture needles (0.20mm diameter, 15mm length) on each of the identified acupuncture points (Shen men, Point zero, brain, thalamus, Pineal, Master cerebral, Insomnia 1, Kidney, Heart, Insomnia 2, Occiput, Forehead) to bilateral ears for a total of 30 minutes. Acupuncture will be administered by a board certified Psychiatrist with supplemental privileges to perform acupuncture.
  Arms: Auricular Acupuncture

SUMMARY:
Post traumatic stress disorder (PTSD) has emerged as a significant problem among troops returning from combat zones. A majority of these veterans will report difficulty maintaining or initiating sleep. The purpose of this research will be to conduct a prospective, randomized, wait list controlled, small scale feasibility study to examine if the use of an auricular acupuncture regimen improves quality of sleep for Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF)veterans with PTSD receiving standard PTSD treatment. Hypothesis: Objective and subjective sleep disturbances and sleep quality will be improved in OIF/OEF veterans who receive auricular acupuncture in conjunction with standard PTSD therapy or standard therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Male gender
* veteran of OIF/OEF
* comorbid mental health problems such as depression, anxiety are allowed
* self-reported sleep disturbance (defined as having one or more of the following-sleep onset latency greater than 30 minutes, two or more awakenings per night, total sleep time less than six hours per night, presence of nightmares.
* sleep disturbances must have started after a deployment

Exclusion Criteria:

* Axis I mental disorders incompatible with active military service
* History of moderate to severe traumatic brain injury
* Sleep Apnea
* Current use of Continuous Positive Airway Pressure Devices
* Significant Co-morbid conditions (heart, lung, liver disease, etc.)
* Other treatment programs that involve cognitive processing therapy
* No concurrent use of acupuncture during study
* taking any anticoagulation medication
* essential tremors

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Objective Sleep Times | Baseline (upon entering study) and at one month
  Change in sleep times will be measured by actigraphy for seven days at baseline and again for seven days at one month.
Change in Subjective Sleep Times | Baseline (upon entering study) and at one month
  Change in subjective sleep times will be measured by sleep diary for one week at baseline and again for seven days at one month
Acceptability of Acupuncture as a Treatment for Sleep Disturbance | One month
  Acceptability of Acupuncture as a treatment for sleep disturbance will be measured at one month by a likert type question.

SECONDARY OUTCOMES:
Change in Sleep Quality | Baseline (upon entering study) and at one month
  Change in sleep quality will be measured by Pittsburgh Sleep Quality Index Scores at baseline and at one month
Change in Sleep Quality | Baseline (upon entering study) and at one month
  Change in sleep quality ratings will also be measured by the consensus sleep diary sleep quality ratings at baseline and at one month.
Change in Depression | Baseline (upon entering study) and at week 3 & at week 5
  Change in depression will be measured by Patient Health Questionnaire, version 9 (PHQ-9) scores at baseline, at week 3, and at week 5.
Change in Post Traumatic Stress Disorder Symptoms | Baseline (upon enterning the study) and week 3 & at week 5
  Change in Post Traumatic Stress Disorder Symptoms will be measured by the Post Traumatic Stress Disorder Checklist at baseline, at week 3, and at week 5.

OTHER OUTCOMES:
Subjects Feedback on Study | Week 5
  An open ended question will examine subject feedback regarding this study.

CONTACTS AND LOCATIONS:
Overall Officials: Heather C King, MSN, Principal Investigator — Naval Medical Center San Diego/ University of San Diego
Locations (1):
- Overcoming Adversity and Stress and Injury Support Clinic, San Diego, California, United States